CLINICAL TRIAL: NCT05297981
Title: Ultrasound Guided Quadratus Lumborum Block Versus Ultrasound Guided Erector Spinae Plane Block for Postoperative Analgesia in Laparoscopic Abdominal Surgeries
Brief Title: Quadratus Lumborum Block Versus Erector Spinae Plane Block for Postoperative Analgesia in Laparoscopic Surgeries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FMASU R 198\2021
Record Dates: First submitted 2022-02-16; First posted 2022-03-28 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-02

CONDITIONS: Postoperative Pain
Keywords: Laparoscopic surgeries; Erector spinae plane block; Quadratus lumborum block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: This randomized prospective study will be carried out in Ain shams university hospitals for 6 months on 82 adult patients with American Society of Anesthesiologists (ASA) Physical Status Class I and II, aged between 30 and 60 years, and scheduled for laparoscopic abdominal surgery after approval by local ethical committee. Written and informed consent will be taken from each patient. Every patient will receive an explanation to the purpose of the study and will have a secret code number to ensure privacy to participant and confidentiality of data.
  Patients will be randomly allocated into two equal groups:
  * Group E (41 patients): Each patient will receive general anesthesia plus bilateral ESP block.
  * Group Q (41 patients): Each patient will receive general anesthesia plus bilateral posterior QLB.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group E (Experimental): Erector spinae plane block
  Interventions: Procedure: Erector spinae plane block
- Group Q (Experimental): Quadratus lumborum block
  Interventions: Procedure: Quadratus lumborum block

INTERVENTIONS:
Procedure: Erector spinae plane block — The patient will be placed in lateral decubitus position. A high frequency linear probe of a transportable Fuji M-Turbo ultrasound system will be placed on the spinous process at T8 level on the parasagittal plane and then slide 2.5-3 cm laterally to visualize the transverse process and erector spinae muscle. Using the inplane technique,then 0.5 ml/kg of 0.25% bupivacaine will be injected between the muscle and transverse process. The same procedure will be performed bilaterally.
  Arms: Group E
Procedure: Quadratus lumborum block — The patient will be placed in the lateral decubitus position. A low frequency curved probe of a transportable Fuji M-Turbo ultrasound system will be placed horizontally in the anterior axillary line midway between the subcostal margin and the iliac crest to identify the triple abdominal muscle layers.A 22-G, 80-mm needle echogenic needle will be inserted in plane relative to the US probe, into the posterior aspect of the QL muscle (between QL and erector spinae muscle); this is known as QLB type 2. Then, 0.5 ml/kg of 0.25% bupivacaine will be injected behind the muscle as a bolus dose. The block will be performed bilaterally.
  Arms: Group Q

SUMMARY:
Postoperative pain after laparoscopic abdominal surgeries can be severe. Despite multimodal analgesia protocols, administration of high doses of opioids is often required hindering early mobilization and discharge of the patient from the day surgery setting and is suboptimal in an Early Recovery after Surgery setting.

Settings and design A prospective randomized double blinded study.

Aim To evaluate and compare the analgesic effect of ultrasound-guided erector spinae plane (ESP) block with ultrasound-guided posterior Quadratus Lumborum Block in laparoscopic abdominal surgeries.

Patients and methods This randomized prospective study will be carried for 6 months on adult patients with American Society of Anesthesiologists (ASA) Physical Status Class I and II, aged between 30 and 60 years.

DETAILED DESCRIPTION:
The role of regional anaesthesia is well established in abdominal surgery, with epidural analgesia being the gold standard in perioperative analgesia since the early 1900s.However early mobilization, minimally invasive surgical techniques, and pharmacologic venous thromboprophylaxis are now recognized as key components of efficient surgical recovery. The search for motor-sparing, less-invasive, safer, and efficacious alternatives to epidural analgesia has been prioritized.

With the introduction of the ultrasound machine in the operating theatres, the practice of regional anaesthesia has been changed from landmark-based techniques to regional blocks administered under direct vision through the ultrasound machine. The ultrasound-guided Erector Spinae Plane (ESP) block is a novel truncal interfacial regional technique.

Two variations of the ESP block for thoracic and abdominal procedures have recently been described in literature. The injection site is either at the level of T5 transverse process, resulting in spread between the C7 and T8 segmental levels, or at the levels of the T7-T9 transverse processes, resulting in spread between the T6 and T12 segmental levels. Quadratus lumborum block (QLB) is a posterior extension of the TAP block. It was first described by Dr Blanco, and it was later modified by Sauter et al. These blocks target both somatic structures covering the anterior abdominal wall, with suggestions of abdominal visceral coverage as well, most commonly using a lateral, posterior, or anterior approach.

The lateral approach (previously QL1) involves depositing local anaesthesia at the lateral border of the QL muscle, anterior to the aponeurosis of the transversus abdominis muscle and within the anterior thoracolumbar fascia. The posterior approach (previously QL2) involves injecting posterior to the QL muscle, in the middle thoracolumbar fascia. The anterior approach (also called the transmuscular (QL block) involves injecting anterior to the QL muscle, between it and the psoas major muscle and in the anterior thoracolumbar fascia.

Patients and Methods

This randomized prospective study will be carried out in Ain shams university hospitals for 6 months on adult patients with American Society of Anesthesiologists (ASA) Physical Status Class I and II, aged between 30 and 60 years, and scheduled for laparoscopic abdominal surgery after approval by local ethical committee. Written and informed consent will be taken from each patient. Every patient will receive an explanation to the purpose of the study and will have a secret code number to ensure privacy to participant and confidentiality of data.

Randomization A computer system will be used for randomization by creating a list of number each number referred to one of the two groups. Block randomization will be used to ensure equality of the groups. Each number will be sealed in an opaque envelope. Then, each patient will be asked to choose one of the envelopes and give to an anesthesiologist who will compare it to the computer-generated list and hence assigned to one of the two groups.

Blinding The patients and the investigators who will be responsible for assessing the primary and secondary outcomes will be blinded to study group assignment. However, the attending intraoperative anaesthesiologists and assessors will not be blinded to study group assignment.

All patients will be assessed preoperatively, and will be instructed to fast for 8 hrs. On arrival to the operation theatre, Intravenous access will be established, and lactated Ringer solution will be infused by rate 10 ml/kg. Patients will receive titration of 0.03 mg/kg midazolam intravenously as sedation. Standard monitors including non-invasive blood pressure, electrocardiogram (ECG), and pulse oximetry (SpO2) and capnography will be applied to monitor the perioperative hemodynamic parameters. For both groups, general anesthesia will be induced with IV injection of fentanyl (1 μg/kg) and propofol (2 mg/kg), and then, atracurium (0.5 mg/kg) will be injected for endotracheal intubation. Mechanical ventilation will be maintained to keep the end-expiratory CO2 values between 34 and 36 mmHg. Anesthesia will be continued with isoflurane 1%-2% in 100% O2. Incremental dose of atracurium (0.1 mg/kg) will be given every 30 min or when needed.

After endotracheal intubation and before the start of the surgery, anesthesiologist will perform the block techniques and will administer the medication. Both blocks will be performed under complete aseptic precautions using ultrasound machine.

In group Q:

The patient will be placed in the lateral decubitus position. After sterilization of the US site, needle entry, and draping, a low frequency curved probe of a transportable Fuji M-Turbo ultrasound system will be placed horizontally in the anterior axillary line midway between the subcostal margin and the iliac crest to identify the triple abdominal muscle layers. Then, the probe will move posteriorly to the posterior axillary line until the QL muscle was appears with its attachment to the lateral edge of the transverse process of the L4 vertebral body, the psoas major muscle anteriorly, and the erector spinae muscle posteriorly; this is a well-recognizable pattern of a shamrock sign with three leaves7. A 22-G, 80-mm needle echogenic needle will be inserted in plane relative to the US probe, into the posterior aspect of the QL muscle (between QL and erector spinae muscle); this is known as QLB type 2. Then, 0.5 ml/kg of 0.25% bupivacaine will be injected behind the muscle as a bolus dose. The block will be performed bilaterally.

In group E:

The patient will be placed in lateral decubitus position. After sterilization of the US site, needle entry, and draping, a high frequency linear probe of a transportable Fuji M-Turbo ultrasound system will be placed on the spinous process at T8 level on the parasagittal plane and then slide 2.5-3 cm laterally to visualize the transverse process and erector spinae muscle. Using the inplane technique, A 22-G, 80-mm needle echogenic needle will be inserted between the transverse process and erector spinae muscle. Then 0.5 ml/kg of 0.25% bupivacaine will be injected between the muscle and transverse process. The same procedure will be performed bilaterally.

Intravenous fentanyl (0.5 µg/kg) will be given intraoperatively when any increase in MAP or HR more than 20% of baseline data occurred throughout the procedure. At the end of the surgery, anesthesia will be discontinued, reversal of muscle relaxation by 0.02 mg/kg atropine and 0.05 mg/kg prostigmine will be given.

Patients will be assessed in the immediate postoperative period and then at 2, 6,12 and at 24 h for the quality of analgesia using Visual analogue scale (VAS) score, and VAS more than 5 will be managed by fixing paracetamol (10 mg/kg) IV every 8 hours and injection of 50 mg of pethidine intravenous as second rescue analgesia.

Primary and Secondary outcomes

The primary outcome of the study The first time to rescue analgesia (recorded within the first 24 hour postoperatively) The time to ask for postoperative analgesia is the time from the end of operation to patient reporting VAS ≥ 5. Pain assessments are conducted by a researcher who is unaware of the grouping.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included in the study aged 30-60 years.
* ASA Physical Status Class I and II.
* Elective laparoscopic abdominal surgery under general anesthesia.

Exclusion Criteria:

* Infection at injection site.
* History of allergy to local anesthetics.
* Coagulation disorders.
* Physical or mental diseases which may interfere with the evaluation of pain scores.
* Kidney failure or liver cell failure.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Estimated)
Dates: Start 2021-11-23 (Actual); Primary Completion 2022-05-10 (Estimated); Study Completion 2022-05-23 (Estimated)

PRIMARY OUTCOMES:
The first time to rescue analgesia | (recorded within the first 24 hour postoperatively)
  The time to ask for postoperative analgesia is the time from the end of operation to patient reporting Visual analogue scale ≥ 5. Pain assessments are conducted by a researcher who is unaware of the grouping

SECONDARY OUTCOMES:
Visual analogue scale (VAS) | measured immediate after surgery, 2,6,12,24 hours postoperatively
  On a scale of 0-10, the patient will learn to quantify postoperative pain where 0= No pain and 10= Maximum worst pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abdelrahman Mohamed, Cairo, Egypt

REFERENCES:
- [Background] 1. Ljungqvist O, Scott M, Fearon KC. Enhanced recovery after surgery: a review. JAMA Surg.2017;152(3):292-298. 2. Hebbard P, Fujiwara Y, Shibata Y, Royse C. Ultrasound-guided transversus abdominis plane (TAP) block. Anaesth Intensive Care. 2007; 35:616-7. 3. M. Forero, S. D. Adhikary, H. Lopez, C. Tsui, and K. J. Chin, "The erector spinae plane block a novel analgesic technique in thoracic neuropathic pain," Regional Anesthesia and Pain Medicine, vol. 41, no. 5, pp. 621-627, 2016. 4. K. J. Chin, S. Adhikary, N. Sarwani, and M. Forero, "The analgesic efficacy of pre-operative bilateral erector spinae plane (ESP) blocks in patients having ventral hernia repair," Anaesthesia, vol. 72, no. 4, pp. 452-460, 2017 5. Sauter AR, Ullensvang K, Niemi G, Lorentzen HT, Bendtsen TF, Børglum J, et al. The Shamrock lumbar plexus block: A dose-finding study. Eur J Anaesthesiol. 2015; 32:764- 70 6. El-Boghdadly K, Elsharkawy H, Short A, Chin KJ. Quadratus lumborum block nomenclature and anatomical considerations. Reg Anesth Pain Med.2016;41(4):548-549 7. Ueshima H, Otake H, Jui-An L. Ultrasound-guided quadratus lumborum block: an updated review of anatomy and techniques. Biomed Res Int. 2017; 2017:1-7 8. Aditianingsih D, Pryambodho AN, Tantri AR, et al. A randomized controlled trial on analgesic effect of repeated quadratus lumborum block versus continuous epidural analgesia following laparoscopic nephrectomy. BMC Anesthesiol. 2019; 19:221 9. Niraj G, Tariq Z. Continuous erector spinae plane (ESP) analgesia in different open abdominal surgical procedures: a case series. J Anesth Surg. 2018;5(1):57-60